CLINICAL TRIAL: NCT05813444
Title: Gingival Phenotype Prevalence of Lower Incisors and Associated Risk Factors in French Dental Students Population : a Cross-sectional Study
Brief Title: Gingival Phenotype Prevalence of Lower Incisors and Associated Risk Factors : a Cross-sectional Study
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Other Study IDs: 23Odonto02
Record Dates: First submitted 2023-04-03; First posted 2023-04-14 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2023-03

CONDITIONS: Gingival Diseases
MeSH Terms: conditions — Gingival Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Main Cohort: Dental students on the university hospital of Nice

SUMMARY:
Several types of gingival phenotype can be diagnosed in the general population and their evaluation is an essential clinical criterion in periodontal practice, whether the periodontal therapies are preventive or curative, non-surgical or surgical. Moreover, several authors have shown that the gingival phenotype varies from one dental sector to another, hence the interest of a meticulous and targeted diagnostic approach in relation to the established therapeutic objectives. To date, the gingival phenotype has been not studied extensively in the mandibular incisal area. Therefore, it seems relevant to conduct an observational cross-sectional study on a cohort of patients in good general health and with a healthy and intact periodontium to assess the prevalence of the gingival phenotype in this area. The secondary objective is to highlight the associated intrinsic and extrinsic risk factors for thin gingival phenotype, to anticipate a risk of gingival recession and to propose an early personal therapy.

ELIGIBILITY:
Inclusion Criteria:

* age (18 years old or older)
* dental student on the university hospital of Nice
* social security affiliate
* systemically healthy
* healthy and intact periodontium
* informed consent.

Exclusion Criteria:

* pregnancy
* under any regular medical treatment
* active periodontal disease
* presence of plaque
* enduring orthodontic treatment
* periodontal surgery in the mandibulary anterior region
* non consent patient
* patient under judgment trials.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Dental student with healthy and intact periodontium
Sampling Method: Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2022-06-29 (Actual); Primary Completion 2023-12-29 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Gingival phenotype prevalence | 18 months
  Assessment of gingival thickness (Kan et al 2015) and keratinised tissue height of the lower incisors with UNC-15 periodontal probe (Hu-Freidy, USA) and clinical photography.

SECONDARY OUTCOMES:
Associated risk factors for thin gingival phenotype | 18 months
  Age, gender, smoking habit, orthodontic background, oral hygiene habit, oral ventilation, dysfunction, facial typology, chin shape, visibility of vascularisation and root convexity through the gum, gingival recession (Cairo), frenal insertion and skin type.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Nice, Nice, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dridi SM, Ameline C, Masucci C, Fontas E, Charavet C. Gingival phenotype prevalence of lower incisors and associated risk indicators in the French dental student population: a cross-sectional study. Clin Oral Investig. 2025 Feb 15;29(2):130. doi: 10.1007/s00784-025-06206-7. PMID 39953292